CLINICAL TRIAL: NCT02550223
Title: Ultrasound Guided Radial Artery Cathetrization, A Novel Technique.
Brief Title: Ultrasound Guided Radial Artery Catheterization
Acronym: US radial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Refa 5
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Arterial Catheterization, Peripheral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oblique (Experimental): Ultrasound guided radial artery catheterization using oblique view obtained by tilting the US probe 30-45 degrees over the course of the artery
  Interventions: Procedure: radial artery Catheterization
- Transverse group (Active Comparator): Ultrasound guided radial artery catheterization using transverse view
  Interventions: Procedure: radial artery Catheterization
- Longitudinal group (Active Comparator): Ultrasound guided radial artery catheterization using longitudinal view
  Interventions: Procedure: radial artery Catheterization

INTERVENTIONS:
Procedure: radial artery Catheterization — Insertion of radial artery catheter for sampling and blood pressure measurement

SUMMARY:
Comparing an novel technique ( oblique view) during ultrasound guided radial artery catheterization versus Transverse and longitudinal views

ELIGIBILITY:
Inclusion Criteria:

* all patients with clear indication to radial artery catheterization like hemodynamic instability or the need of frequent arterial samples

Exclusion Criteria:

* refusal, Peripheral arterial diseases

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
success rate of radial artery cathertrization | postoperate 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140